CLINICAL TRIAL: NCT03577015
Title: International Prospective Registry for the Diagnosis and Management of Disseminated Intravascular Coagulation in the Intensive Care Unit
Brief Title: International Prospective Registry of Disseminated Intravascular Coagulation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marcella Muller (Other)
Collaborators: Università degli Studi dell'Insubria (Other); University of Chieti (Other); Ospedale S. Antonio (Unknown); Poliambulanza Foundation Hospital (Unknown); Manchester Royal Infirmary (Unknown); Juntendo University (Other)
Responsible Party: Sponsor-Investigator, Marcella Muller, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Other Study IDs: 184/2017
Record Dates: First submitted 2018-05-22; First posted 2018-07-05 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Disseminated Intravascular Coagulation
Keywords: disseminated intravascular coagulation; sepsis; trauma; pancreatitis; malignancy; obstetric complication
MeSH Terms: conditions — Disseminated Intravascular Coagulation; Sepsis; Wounds and Injuries; Pancreatitis; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- critically ill patients at risk for DIC: patients 18 years or older with a condition potentially associated with DIC, admitted to intensive care: severe infection/sepsis, solid tumor, hematologic malignancies, trauma, obstetric complications, acute pancreatitis

SUMMARY:
Objectives: to evaluate the current diagnostic and therapeutic approaches for sepis-associated disseminated intravascular coagulation (DIC) in a large prospective registry.

Design: prospective, multicenter, international registry. Study population: patients 18 years or older with severe infection to be potentially associated with DIC will be eligible for the study. The clinical visits and monitoring of the patients will follow local routine practices. No specific imaging tests or laboratory evaluations will be required and patients will be evaluated and treated according to local policy. All the involved centers will be asked to update information on included patients at 2, 4, 6, 8, 10 and 28 days after severe infection diagnosis.

Study outcomes: The primary outcome of the study is the development of DIC. Secondary outcomes are thrombotic (arterial and venous) and bleeding events, overall mortality at 28 days.

Study sample, feasibility, and analysis plan: We plan to enroll a minimum of 1000 patients.

ELIGIBILITY:
Inclusion Criteria:

* admission to the intensive care unit
* 18 years or older

AND one of the following conditions:

* sepsis/severe infection
* solid tumor
* hematological malignancy
* trauma
* obstetric complications
* acute pancreatitis

Exclusion Criteria:

-<18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients 18 years or older with a condition potentially associated with DIC, admitted to the intensive care unit, will be eligible for the study. The maximal time-window allowed between the diagnosis of the disease and inclusion in the study will be 72 hours.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
disseminated intravascular coagulation | 28 days
  occurence of disseminated intravascular coagulation:
  International Society Thrombosis Hemostasis DIC score >4 points (range 0-8 points) items scored: platelet count, prothrombin time, fibrinogen related marker, fibrinogen level
  Japanese Association for Acute Medicine DIC score >3 points (range 0-8)points items scored: inflammatory response, platelet count, prothrombin time, fibrinogen degradation products
disseminated intravascular coagulation | 28 days
  occurence of disseminated intravascular coagulation:
  Japanese Association for Acute Medicine DIC score >3 points (range 0-8)points items scored: inflammatory response, platelet count, prothrombin time, fibrinogen degradation products

SECONDARY OUTCOMES:
mortality | 28 days
  mortality rates in patient who develop or do not develop disseminated intravascular coagulation
venous thromboembolic events | 28 days
  occurence of symptomatic venous thromboembolic events including pulmonary embolism and deep vein thrombosis (VTE) of the upper and lower limbs, visceral VTE, and cerebral VTE.
Arterial thromboembolic events | 28 days
  occurence of arterial thromboembolic events including myocardial infarction, stroke, peripheral embolism
Major and clinically-relevant non-major bleeding | 28 days
  occurence of major and clinically relevant non-major bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Boraso, MD, Principal Investigator — OSPEDALE S. ANTONIO, Padova, Italy; Marcello Di Nisio, MD PhD, Principal Investigator — University of Chieti, Italy; Jecko Tachil, MD PhD, Principal Investigator — Manchester Royal Infirmary, Manchester, England; Pierluigi Ferretti, MD, Principal Investigator — Fondazione Poliambulanza, Brescia, Italy; Toshiaki Iba, MD PhD, Principal Investigator — (Juntendo University, Department of Emergency and Disaster Medicine, Tokyo, Japan
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands